CLINICAL TRIAL: NCT03052634
Title: A Phase Ib Study to Evaluate the Efficacy, Safety and Pharmacokinetics of RC48-ADC for Injection in Subjects With Advanced Breast Cancer With HER2 Positive or HER2 Low Expression
Brief Title: A Study of RC48-ADC in Subjects With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C003 CANCER
Record Dates: First submitted 2017-01-04; First posted 2017-02-14 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2022-01

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RC48-ADC 1.5 mg/kg (HER2 Positive) (Experimental)
  Interventions: Drug: RC48-ADC 1.5 mg/kg (HER2 Positive)
- RC48-ADC 2.0 mg/kg (HER2 Positive) (Experimental)
  Interventions: Drug: RC48-ADC 2.0 mg/kg (HER2 Positive)
- RC48-ADC 2.5 mg/kg (HER2 Positive) (Experimental)
  Interventions: Drug: RC48-ADC 2.5 mg/kg (HER2 Positive)
- RC48-ADC 2.0 mg/kg (HER2 Low Expression) (Experimental)
  Interventions: Drug: RC48-ADC 2.0 mg/kg (HER2 Low Expression)

INTERVENTIONS:
Drug: RC48-ADC 1.5 mg/kg (HER2 Positive) — 15 advanced breast cancer participants with HER2 Positive will be treated with RC48-ADC at a dose of 1.5 mg/kg, every 2 weeks. They will continue the medication until one of the following conditions occurred: disease progression, intolerance of toxicity, withdrawal of informed consent, or treatment for 1 year.
  Arms: RC48-ADC 1.5 mg/kg (HER2 Positive)
Drug: RC48-ADC 2.0 mg/kg (HER2 Positive) — 15 advanced breast cancer participants with HER2 Positive will be treated with RC48-ADC at a dose of 2.0mg/kg, every 2 weeks. They will continue the medication until one of the following conditions occurred: disease progression, intolerance of toxicity, withdrawal of informed consent, or treatment for 1 year.
  Arms: RC48-ADC 2.0 mg/kg (HER2 Positive)
Drug: RC48-ADC 2.5 mg/kg (HER2 Positive) — 15 advanced breast cancer participants with HER2 Positive will be treated with RC48-ADC at a dose of 2.5 mg/kg, every 2 weeks. They will continue the medication until one of the following conditions occurred: disease progression, intolerance of toxicity, withdrawal of informed consent, or treatment for 1 year.
  Arms: RC48-ADC 2.5 mg/kg (HER2 Positive)
Drug: RC48-ADC 2.0 mg/kg (HER2 Low Expression) — 45 advanced breast cancer participants with HER2 Low Expression will be treated with RC48-ADC at a dose of 2.0 mg/kg, every 2 weeks. They will continue the medication until one of the following conditions occurred: disease progression, intolerance of toxicity, withdrawal of informed consent, or treatment for 1 year.
  Arms: RC48-ADC 2.0 mg/kg (HER2 Low Expression)

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics of RC48-ADC for injection in subjects with advanced breast cancer with HER2 positive or HER2 low expression

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed informed consent;
2. Female, aged between 18 to 70 years;
3. ECOG performance status score of 0 or 1;
4. Life expectancy greater than 12 weeks；
5. Patients with locally advanced or metastatic breast cancer diagnosed by histology or cytology, and:

   1. Core cohort: standard treatment is ineffective (the disease progresses or has no remission after treatment) or cannot tolerate standard treatment, or HER2 positive who cannot receive standard treatment (immunohistochemistry is 2+ and confirmed by fluorescence in situ hybridization [FISH] Positive, or immunohistochemical 3+) patients;
   2. Explorative cohort:standard treatment is ineffective (the disease progresses or has no remission after treatment) or cannot tolerate standard treatment, or had no optional standard treatment for HER2 immunohistochemistry 2+ with FISH negative or HER2 immunohistochemistry 1+ (FISH negative or untested). Subjects in the explorative cohort can provide HER2 detection of tumor primary or metastatic site specimens;
6. Measurable lesion according to the RECIST 1.1;
7. Adequate organ function:

(1)absolute neutrophil count(ANC) >= 1.5 x 10(9)/L; (2) platelets>=100*10(9)/L; (3)Total serum bilirubin <=1.5*ULN; (4)serum aspartate transaminase (AST）and serum alanine transaminase (ALT) <=2.5*ULN, or AST and ALT<=5*ULN with hepatic metastasis; (5) Serum creatinine clearance rate >= 45 mL/min; (6) INR<=1.5*ULN and APTT<=1.5*ULN; 8.Women of child-bearing potential and men must agree to use adequate contraception (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices, complete sexual abstinence, or sterilized partner) prior to study entry and during the period of therapy and for 6 months after the last dose of study drug; 9.Left ventricular ejection fraction (LVEF) >= 50%.

Exclusion Criteria:

1. Women who are pregnant (positive blood test before medication) or breastfeeding;
2. Patients received anti-cancer therapy within 4 weeks before study drug treatment;, including chemotherapy, radiotherapy, surgery or hormone therapy, molecular targeted therapy (including trastuzumab etc.); Using Trastuzumab emtansine(T-DM1) or participating in the clinical trial on ADC drugs targeting HER2 and bispecific antibodies targeting HER2;
3. The patient have third interstitial fluid (a large number of pleural effusion or ascites) which has clinical symptom or can not be controlled by drainage or other methods;
4. Received Palliative radiation therapy for bone metastases within 2 weeks before study drug treatment;
5. Toxicity of previous anti-tumor treatment has not recovered to CTCAE [version 4.0] 0-1, except for hair loss;
6. Participated in other clinical trials within 4 weeks;
7. Known hypersensitivity or delayed hypersensitivity to the some components of RC48-ADC or similar drugs;
8. The active infection with clinical significance according to the researcher's judgment;
9. Diagnosed with HBsAg or HBcAb positive and HBV DNA positive, or HCV Ab positive, or HIV Ab positive.
10. Have a history of immunodeficiency, including a positive HIV test, or other acquired, congenital immunity Epidemic defects, or a history of organ transplantation;
11. Uncontrolled systemic diseases such as diabetes, hypertension, Pulmonary fibrosis, acute lung disease, interstitial lung disease, etc.
12. Congestive heart failure with grade 2 or higher (including grade 2) of the New York Institute of Cardiology (NYHA) of the United States in the history of diseases such as acute myocardial infarction, unstable angina, stroke, or transient ischemic attack within 6 months prior to entry ;
13. Insufficient adherence to participate in this clinical study;
14. Patients who had received systemic steroid therapy for a long time(Patients who had received systemic steroid therapy for short time and stopped drug more than 2 weeks could be enrolled );
15. Primary brain or metastatic tumor;
16. Peripheral neuropathy with grade≥2;
17. People with a history of mental illness that is difficult to control.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-12-23 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
RP2D | Estimated 2 year
  Recommended Phase II Dose

SECONDARY OUTCOMES:
Cmax | Estimated 2 year
  Maximum Observed Plasma Concentration
AUC | Estimated 2 year
  Area Under Curve
Tmax | Estimated 2 year
  Time for Cmax
Overall response Rate (ORR) | Estimated 2 year
  As per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 - to estimate the anti-tumor activity of RC48-ADC.
Clinical Benefit Rate (CBR) | Estimated 2 year
  Clinical Benefit Rate was defined as the percentage of patients with complete remission (CR) partial remission (PR) stable (SD) not less than 4 months.
Progression Free Survival (PFS) | Estimated 2 year
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Study Director — RemeGen Co., Ltd.
Locations (7):
- China (7):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The first bethune hospital of jilin unversity, Changchun, Jilin
  - Liaoning cancer hospital & institute, Shenyang, Liaoning
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - Affiliated cancer hospital of Harbin medical university, Harbin
  - The fourth hospital of Hebei medical university, Hebei
  - Jiangsu Cancer Hospital, Nanjing

IPD SHARING:
Plan to Share IPD: No